CLINICAL TRIAL: NCT03251066
Title: Open, Not Randomised, Non-blinded Observation Study to Investigate the Immediate Effect of Proponent - Nasal - Spray in Case of Unspecific Discomfort in the Nose
Brief Title: Immediate Effect of Proponent-Nasal-Spray on Unspecific Discomfort in the Nose
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PRECLIN Biosystems AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PNSY2
Record Dates: First submitted 2017-08-07; First posted 2017-08-16 (Actual); Last update posted 2017-08-21 (Actual); Status verified 2017-08

CONDITIONS: Unspecified Disorder of Nose and Nasal Sinuses
Keywords: Nose Saline Solution Irrigation Nasal Spray; Sodium propionate Locke-Ringer Solution

STUDY DESIGN:
Intervention Model Description: Every participant of the study will specify at the beginning of the investigation his subjective starting situation concerning the nasal discomfort.The participant records his/ her personal impression on the change of severity of the general symptoms or selected individual symptoms of unspecific nasal discomfort following the single administration of "Proponent Nasal Spray". Every Patient serves as his own control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Test group (Other): Proponent Nasal Spray Medical device
  Interventions: Other: Proponent Nasal Spray

INTERVENTIONS:
Other: Proponent Nasal Spray — The medical device consists of a Saline solution containing sodium propionate which is administered as single dose

SUMMARY:
Investigation of the immediate effect on subjective relief of symptoms by Proponent - Nasal - Spray after a one time administration (following a single dose administration in each nostril) in an open, not randomised, non-blinded single centre observation study on 40 volunteers between 18-75 years of age with an unspecific discomfort in the nose such as enhanced nasal discharge/ secretion (runny nose), congested nose, sneezing, itchy nose or feeling of a dry nose.

DETAILED DESCRIPTION:
By regularisation of environment of nasal mucosa and the following restitution and improvement of the ciliary function the efficacy of mucociliary clearance can be remarkably enhanced, pathogens from the environment can be physically removed and a bacterial or viral infection may be prevented on this way.

Such an optimizing effect may be reached by the administration of an equilibrated saline solution with an optimal composition regarding osmolality, pH-value and buffer substance.

In addition it would be very advantageous to support the efficacy of the local unspecific and specific immune mechanisms in the nasal respiratory mucosa (NALT) without any negative effects on the optimized mucociliary clearance.

As demonstrated recently in airway mucosa sodium propionate is able to interact with macrophages, the interleukin system and other factors of the TNF receptor family.

Sodium propionate could therefore have an ancillary effect on the genuine immune mechanisms of nasal respiratory mucosa. On this way the primary effect of administration of saline solution is supported.

ELIGIBILITY:
Inclusion Criteria:

Key inclusion criteria are one or more of the following symptoms:

* nasal discharge/ secretion (runny nose)
* congested nose
* sneezing
* itchy nose
* feeling of a dry nose

Exclusion Criteria:

Key exclusion criteria:

* <18 years of age
* 75 years of age

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2017-04-27 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the safety endpoint (adverse events non-response rate). | up to 48 hrs
  This endpont is defined by the adverse events non-response rate based on the individual adverse events reported by the participant up to 60 min after treatment. The adverse events are specified and defined by scores. The sum score over time for all individual adverse event symptoms will be determined for each participant. Not more than 10 % of all participants of the study should report adverse events with a sum score > 3 for one or more of the listed adverse events. Not more than 10 % of all participants of the study should report adverse events with a sum score > 3 for one or more of the listed adverse effects.

SECONDARY OUTCOMES:
The secondary endpoints of the study are the immediate response rate based on the "Change of severity of general and selected individual symptoms of unspecific nasal discomfort". | up to 48 hrs
  The first co-secondary endpoint of the study is the immediate response rate based on the "Change of severity of general symptoms of unspecific nasal discomfort" following the single administration of "Proponent Nasal Spray" up to 60 min after treatment. The second co-secondary endpoint is the immediate response rate based on the "Change of severity of selected individual symptoms" of nasal discomfort following the single administration of "Proponent Nasal Spray" up to 60 min after treatment - provided the respective symptom was identified by a participant prior to the administration of "Proponent Nasal Spray" as a nasal discomfort.

CONTACTS AND LOCATIONS:
Overall Officials: Soyka Michael, MD, Principal Investigator — ORL, USZ
Locations (1):
- Klinik für Ohren-, Nasen-, Hals- und Gesichtschirurgie University Zürich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Trompette A, Gollwitzer ES, Yadava K, Sichelstiel AK, Sprenger N, Ngom-Bru C, Blanchard C, Junt T, Nicod LP, Harris NL, Marsland BJ. Gut microbiota metabolism of dietary fiber influences allergic airway disease and hematopoiesis. Nat Med. 2014 Feb;20(2):159-66. doi: 10.1038/nm.3444. Epub 2014 Jan 5. PMID 24390308
- [Result] Brandtzaeg P. Immune functions of nasopharyngeal lymphoid tissue. Adv Otorhinolaryngol. 2011;72:20-4. doi: 10.1159/000324588. Epub 2011 Aug 18. PMID 21865681
- [Result] Achilles N, Mosges R. Nasal saline irrigations for the symptoms of acute and chronic rhinosinusitis. Curr Allergy Asthma Rep. 2013 Apr;13(2):229-35. doi: 10.1007/s11882-013-0339-y. PMID 23354530